CLINICAL TRIAL: NCT06480695
Title: Effects of Exercise Training Intensity and Inorganic Nitrate Supplementation on Vascular Health and Fitness in Post-Menopausal Females
Brief Title: Exercise Training Intensity and Nitrate Supplementation in Post-Menopausal Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSR231665
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Menopause
Keywords: Inorganic Nitrate; Menopause; High Intensity Exercise; Vascular Health
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one-month of either high or moderate aerobic exercise training and then further randomized to nitrate or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A study team member not associated with the trial will perform the randomization scheme for the supplementation. Exercise groups will not be blinded but data will not be analyzed until the end or re-labeled by another team member so assessors are unaware while analyzing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nitrate-Rich Beetroot Juice + High Intensity Exercise (HIE) (Experimental): Participants assigned to this group will be instructed to consume 1 bottle of nitrate-rich beetroot juice (~400mg of nitrate each) 2x a day (morning a night) starting 2-hours before the first exercise session. Participants will complete a supervised bout of exercise on a treadmill 3x a week for 1-month. Participants will exercise at an RPE of 15-17 based on the participant's VO2peak test.
  Interventions: Dietary Supplement: Nitrate-Rich Beetroot Juice; Behavioral: High Intensity Exercise
- Nitrate-Depleted Placebo Beetroot Juice + High Intensity Exercise (HIE) (Placebo Comparator): Participants assigned to this group will be instructed to consume 1 bottle of nitrate-depleted beetroot juice 2x a day (morning a night) starting 2-hours before the first exercise session. Participants will complete a supervised bout of exercise on a treadmill 3x a week for 1-month. Participants will exercise at an RPE of 15-17 based on the participant's VO2peak test.
  Interventions: Behavioral: High Intensity Exercise; Dietary Supplement: Nitrate-Depleted Placebo Beetroot Juice
- Nitrate-Rich Beetroot Juice + Moderate Intensity Exercise (MIE) (Active Comparator): Participants assigned to this group will be instructed to consume 1 bottle of nitrate-rich beetroot juice (~400mg of nitrate each) 2x a day (morning a night) starting 2-hours before the first exercise session. Participants will complete a supervised bout of exercise on a treadmill 3x a week for 1-month. Participants will exercise at an RPE of 10-12 based on the participant's VO2peak test.
  Interventions: Dietary Supplement: Nitrate-Rich Beetroot Juice; Behavioral: Moderate Intensity Exercise
- Nitrate-Depleted Placebo Beetroot Juice + Moderate Intensity Exercise (MIE) (Placebo Comparator): Participants assigned to this group will be instructed to consume 1 bottle of nitrate-depleted beetroot juice 2x a day (morning a night) starting 2-hours before the first exercise session. Participants will complete a supervised bout of exercise on a treadmill 3x a week for 1-month. Participants will exercise at an RPE of 10-12 based on the participant's VO2peak test.
  Interventions: Behavioral: Moderate Intensity Exercise; Dietary Supplement: Nitrate-Depleted Placebo Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Nitrate-Rich Beetroot Juice — subjects will consume 1 bottle of nitrate-rich beetroot juice (~400mg of nitrate each) 2x a day
  Other Names: Inorganic Nitrate; James White Beet It
  Arms: Nitrate-Rich Beetroot Juice + High Intensity Exercise (HIE); Nitrate-Rich Beetroot Juice + Moderate Intensity Exercise (MIE)
Behavioral: High Intensity Exercise — exercise at an intensity midway between the lactate threshold and VO2peak, from the screening test at an RPE of ~ 15-17
  Arms: Nitrate-Depleted Placebo Beetroot Juice + High Intensity Exercise (HIE); Nitrate-Rich Beetroot Juice + High Intensity Exercise (HIE)
Behavioral: Moderate Intensity Exercise — exercise at the RPE at LT associated an ~ RPE of 10-12
  Arms: Nitrate-Depleted Placebo Beetroot Juice + Moderate Intensity Exercise (MIE); Nitrate-Rich Beetroot Juice + Moderate Intensity Exercise (MIE)
Dietary Supplement: Nitrate-Depleted Placebo Beetroot Juice — Subjects will consume 1 bottle of nitrate-depleted beetroot juice 2x a day
  Arms: Nitrate-Depleted Placebo Beetroot Juice + High Intensity Exercise (HIE); Nitrate-Depleted Placebo Beetroot Juice + Moderate Intensity Exercise (MIE)

SUMMARY:
Menopause greatly increases cardiovascular disease risk (CVD). Current exercise guidelines are inadequate to ameliorate this risk and higher intensity exercise may be necessary for cardiovascular benefits in postmenopausal females. Oral nitrate supplementation enhances exercise performance and CVD risk profile in several clinical conditions. The investigators recently reported that 3-days of nitrate supplementation in postmenopausal females enhances acute post-exercise vascular function, in an intensity dependent manner. The effects of nitrate supplementation and exercise training over a longer training program remains unexplored. This investigation will examine the impact of exercise training intensity with and without inorganic nitrate supplementation, on CVD and fitness outcomes. Postmenopausal females will be tested for maximal oxygen uptake and lactate threshold before randomization to one of four groups: that inorganic nitrate-rich beetroot juice, or beetroot juice with nitrate extracted; and assigned to one-month of calorie matched high-intensity or moderate-intensity exercise training. Vascular function and fitness will be evaluated before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female (greater than age 45 but less than age 75)
* Sedentary (does not exercise regularly or less than 2 bouts of exercise per week)
* No major changes in medication in the last 3 months

Exclusion Criteria:

* Smokers within last 5 years
* Weight unstable (loss/gain of more than 3kg in the past 3 months)
* Any medical condition that prevents the subject from exercising safely
* Hormone replacement therapy (current or within last 3 months)
* Diabetes
* Currently or recently on vasoactive medications (i.e., calcium channel blockers, statins, ACE or renin inhibitors, ARBs, nitrates, alpha- or beta-blockers, diuretics, proton pump inhibitors, etc.)
* Oral antibiotic use within previous four weeks
* Oral disease or poor oral health as determined by the Oral Health Questionnaire
* Using an antibacterial mouthwash or a mouthwash containing chlorhexidine and unwilling to discontinue use

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Function (Flow-Mediated Dilation [FMD]) | Baseline and after 1-month of exercise training
  Participants will be placed in a supine position with their left forearm slightly extended and supinated with legs straight. The arteries will be imaged using a high-resolution 7.5MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 3 minutes post-occlusion; an EKG trigger will be used to capture images during end-diastole of the cardiac cycle.
Cardiorespiratory Fitness | Baseline and after 1-month of exercise training
  Peak aerobic capacity (VO2peak) will be assessed using a symptom-limited graded exercise test on a treadmill. An IV will be placed and lactate measured during rest and after the completion of every 3-minute stage to determine lactate threshold at VO2peak.

SECONDARY OUTCOMES:
Oral Nitrate Reducing Capacity | Baseline and after 1-month of exercise training
  Assessment of the oral microbiome's ability to reduce nitrate to nitrite. This will be measured through an unstimulated saliva sample and a rinse of a standard nitrate solution.
Skeletal muscle perfusion | Baseline and after 1-month of exercise training
  Skeletal Muscle Blood Flow (straight gauge plethysmography) will be measured non-invasively using venous occlusion/strain-gauge plethysmography both at rest and during reactive hyperemia following 5-minutes of occlusion via the Hokanson A16. A strain gauge device will be place around the widest part of the participant's right calf. A blood pressure place around participant's ankle will be inflated for 60 seconds to eliminate foot circulation from the measurement. At the same time, a cuff placed on the thigh will be inflated to block venous blood flow. The cuff occlusion will be held for ~60 seconds ((several cardiac cycles (4-6 cycles)) to obtain resting blood flow measurements.
Peripheral and Central Blood Pressures | Baseline and after 1-month of exercise training
  Brachial artery blood pressures will be obtained using a standard sphygmomanometer. Aortic blood pressures will be obtained using applanation tonometry (SphygmoCor version 8.0, AtCor Medical).
24-hour ambulatory blood pressure | Baseline and after 1-month of exercise training
  Blood pressure will be monitored using a standard ambulatory brachial artery blood pressure cuff (SunTech Oscar 2, SunTech Medical). Blood pressure measurements are programmed to be taken every 30-minutes during the day and every hour at night. This allows for monitoring of nighttime blood pressure changes and variations throughout the day.
Skeletal muscle microvascular perfusion (near-infra-red- spectroscopy) | Baseline and after 1-month of exercise training
  Tissue oxygenation will be captured noninvasively using non-invasive, near-infrared spectrometry (NIRS, PortaMon, Artinis Medical Systems B.V., The Netherlands) positioned on the gastrocnemius or vastus lateralis muscle.
Lipids | Baseline
  A blood sample will be obtained to measure lipids.
Hemoglobin | Baseline and after 1-month of exercise training
  A blood sample will be obtained to measure hemoglobin.
Plasma Nitrate | Baseline and after 1-month of exercise training
  A fasting blood draw will be taken. Following the blood draw, the participant will take one dose of Beetroot juice. The participant will then return to the lab three hours later for a second blood draw to assess level of nitrate in the plasma.
Plasma Nitrite | Baseline and after 1-month of exercise training
  A fasting blood draw will be taken. Following the blood draw, the participant will take one dose of Beetroot juice. The participant will then return to the lab three hours later for a second blood draw to assess level of nitrite in the plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Allen, PhD, Principal Investigator — UVA
Locations (1):
- Student Health and Wellness Building - Department of Kinesiology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No